CLINICAL TRIAL: NCT01959555
Title: Project to Update the Study of Congenital Haemophilia in Spain
Acronym: PUCHS
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HAEM-4076; U1111-1136-7052 (Other: WHO); NOV-HEM-2013-01 (Other: Novo Nordisk)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrospective collection of data
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Patients will not be treated with any specific product. Data collection only.

SUMMARY:
This study is conducted in Europe. The aim of the study is to update the knowledge about the prevalence and severity of congenital haemophilia (A and B) in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. (Study-related activities are any procedure related to recording of data according to the protocol)
* Male patients of any age diagnosed with congenital haemophilia A or B who visited their HTC at least once during the period of January 2013 to December 2013

Exclusion Criteria:

* Previous participation in this study
* Female patients
* Acquired haemophilia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in active follow-up in HTCs (Haemophilia Treatment Centres) will be included in this study. A patient is considered as active if a visit to the HTC is performed in the period of January 2013 to December 2013.
Sampling Method: Non-Probability Sample
Enrollment: 1157 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of congenital haemophilia A and B in Spain in 2013, described as proportion (%) of patients in the total population (extracted from the last available census of the Spanish population for the regions considered for the study) | Assessed at study visit (day 1)
Severity (mild, moderate or severe) of congenital haemophilia A and B in Spain during 2013, described as proportion (%) per category of the total number of patients with haemophilia A or B | Assessed at study visit (day 1)

SECONDARY OUTCOMES:
Mean current age at the time of visit to the HTC in 2013 | Assessed at study visit (day 1)
Mean age at diagnosis | Assessed at study visit (day 1)
Proportion (%) of patients with/without genetic screening performed | Assessed at study visit (day 1)
Proportion (%) of patients who needed support of a reference Haemophilia Healthcare Centre in 2013 | Assessed at study visit (day 1)
Proportion (%) of patients who received plasmatic or recombinant treatment | Assessed at study visit (day 1)
Proportion (%) of patients who received on demand or prophylaxis treatment | Assessed at study visit (day 1)
Mean number of bleeding episodes | Assessed at study visit (day 1)
Mean number of joint bleeds | Assessed at study visit (day 1)
Proportion (%) of patients with established arthropathy | Assessed at study visit (day 1)
Proportion (%) of patients with infectious complications | Assessed at study visit (day 1)
Proportion (%) of patients with HIV (Human immunodeficiency virus) | Assessed at study visit (day 1)
Proportion (%) of patients with presence of inhibitors | Assessed at study visit (day 1)
Proportion (%) of patients with immune tolerance induction treatment performed | Assessed at study visit (day 1)
Total number of surgery interventions performed | ThAssessed at study visit (day 1)
Proportion (%) of patients with quality of life questionnaire (QoLQ) performed in 2013 | Assessed at study visit (day 1)
Mean number of days of absenteeism to school/university in children and adolescents in 2013 | Assessed at study visit (day 1)
Mean number of days of absenteeism from work in 2013 | Assessed at study visit (day 1)
Proportion (%) of patients with treatment administered at home | Assessed at study visit (day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Madrid, Spain

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com